CLINICAL TRIAL: NCT05090384
Title: Serial Response and Biomarker-Guided Steroid Taper for Children With GVHD
Brief Title: Pediatric GVHD Low Risk Steroid Taper Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Levine (Other)
Responsible Party: Sponsor-Investigator, John Levine, Professor of Internal Medicine and Pediatrics, Director of BMT Clinical Research, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 21-0541
Record Dates: First submitted 2021-10-12; First posted 2021-10-22 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Acute Graft vs Host Disease; Allogeneic Bone Marrow Transplantation; Adverse Effects
Keywords: acute Graft vs Host Disease; aGVHD; Pediatric; steroid taper; MAP; allogeneic hematopoietic stem cell transplantation
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: All enrolled patients start on the same dose of steroids for treatment of GVHD, blood samples are taken at week 1 and 2 post study start and biomarkers plus clinical response determines how steroid treatment is continued
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Steroid Taper (Experimental): All enrolled patients start on the same dose of steroids for treatment of GVHD, blood samples are taken at week 1 and 2 post study start and biomarkers plus clinical response determines how steroid treatment is continued
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Prednisone starting dose of 0.5 mg/kg; for patients who respond clinically and continue to have low biomarkers will be tapered rapidly; those that are not clinically responding or whose biomarkers increase will be treated per their treating physicians plan or by standard of care

SUMMARY:
The standard treatment for acute graft-vs-host disease (GVHD) is to suppress the activity of the donor immune cells using steroid medications such as prednisone. Although most GVHD, especially in children, responds well to treatment, sometimes (around 1/3 of the time) there is either no response to steroids or the response does not last. In those cases, the GVHD can become dangerous and even life-threatening. Unfortunately, doctors cannot predict who will have a good response to treatment based on symptom severity or initial response to steroids. As a result, nearly all children who develop GVHD are treated with long courses of high dose steroids even though that means many patients receive more treatment than they probably need. Steroid treatment can cause short-term complications like infections, high blood sugar, high blood pressure, muscle weakness, depression, anxiety, and problems sleeping and long-term complications like bone damage, cataracts in the eyes, and decreased growth. The risk of these complications increases with higher doses of steroids and longer treatment. It is important to find ways to decrease the steroid treatment in patients who do not need long courses.

The doctors conducting this research have developed a blood test (GVHD biomarkers) that predicts whether a patient will respond well to steroids. The study team found that children who have low GVHD biomarkers at the start of treatment and for the first two weeks of treatment have a very high response rate to steroids. In this study, the study team will monitor GVHD symptoms and biomarkers during treatment and taper steroids quickly in patients who have GVHD that is expected to respond very well to treatment. The study team will assess how many patients respond well to lower steroid dosing and what steroid complications develop. The study team will also use surveys to obtain the patient's own assessment of their quality of life (down to age 5 years).

DETAILED DESCRIPTION:
Pediatric patients with Minnesota standard risk GVHD that is also Ann Arbor 1 by biomarkers will begin treatment at 0.5 mg/kg/d prednisone (or other steroid equivalent). Patients with favorable clinical responses and biomarker scores at weeks 1 and 2 will have their steroid doses tapered quickly on a weekly basis for four weeks. Patients whose GVHD does not respond or have unfavorable biomarker scores will have their steroid doses increased and be removed from study treatment. The primary endpoint is the proportion of patients whose cumulative steroid dose for the first four weeks is less than half of standard dosing.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed GVHD that meets criteria for Minnesota standard risk (see section 9.0) except isolated skin rash <25% body surface area without other manifestations.
* Ann Arbor 1 GVHD by biomarkers
* GVHD not previously treated systemically (topical therapies and non-absorbed steroids are allowed)
* Any donor type, HLA-match, conditioning regimen is acceptable
* Age 0-21 years at the time of screening
* Signed and dated written informed consent obtained from patient or legal representative and assent from pediatric patients capable of providing assent

Exclusion Criteria:

* Patients treated for GVHD with >0.5 mg/kg/day prednisone for any duration or any steroid treatment for GVHD for more than 2 days prior to screening.
* Patients receiving corticosteroids >0.1 mg/kg prednisone (or other steroid equivalent) for any indication within 7 days before the onset of acute GVHD except for adrenal insufficiency, premedication for transfusions/IV medications, or intermittent use for symptom control such as nausea/vomiting
* Relapsed, progressing, or persistent malignancy or other condition (e.g., known declining donor chimerism) requiring withdrawal of systemic immune suppression or donor leukocyte infusion (DLI)
* Patients with uncontrolled infection (i.e., progressive symptoms related to infection despite treatment, persistently positive microbiological cultures despite treatment, viral reactivations unresponsive to treatment, or any other evidence of severe infection)
* A clinical presentation resembling de novo chronic GVHD or overlap syndrome developing before or present at the time of enrollment
* Patients who are pregnant
* Patients requiring mechanical ventilation or cardiac pressor support

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of CR, VGPR, or PR on day 28 with low cumulative steroid exposure | study day 28
  Proportion of patients with low-risk GVHD (Minnesota standard risk/Ann Arbor 1) who are in CR, VGPR or PR on day 28 and whose cumulative prednisone (or other steroid equivalent) exposure during the first four weeks of treatment is ≤13.5 mg/kg and who have had no intervening additional GVHD therapy for those in CR or VGPR.
  Complete Response (CR): All evaluable organs (skin, liver, GI tract) stage 0. Very Good Partial Response (VGPR): Any response that approximates a CR with the exception of rash <25% body surface area.
  Partial Response (PR): An improvement in one or more organ involved with GVHD symptoms without worsening in others.

SECONDARY OUTCOMES:
Treatment response by day 28 | study day 28
  Proportion of patients who achieve a treatment response by day 28 of treatment. Treatment responses are defined as complete response (CR), very good partial response (VGPR), or partial response (PR). For a response to be scored as CR, VGPR, or PR on day 28, the patient must be in response on day 28 and have had no intervening systemic therapy for acute GVHD other than steroids.
Serious infection rate | study day 90
  Proportion of patients who develop serious infections (viral, bacterial, fungal, parasitic as defined in protocol)
  Serious infections are defined using the standardized criteria widely used for clinical trials at academic BMT centers, such as life-threatening fungal infections or hemorrhagic cystitis from BK viral infection and include clinically significant CMV infections that require anti-viral treatment regardless of end-organ damage, given the toxicity of such treatments. Serious infections include any viral, bacterial, fungal or parasitic infections that requires systemic treatment.
Overall survival at 6 months | 6 months
  Overall survival at 6 months
  OS is defined as the time from the first dose of study treatment to the date of death (whatever the cause).
Overall survival at 12 months | 12 months
  Overall survival at 12 months
  OS is defined as the time from the first dose of study treatment to the date of death (whatever the cause).
Cumulative incidence of Non-Relapse Mortality (NRM) at 6 months | 6 months
  Cumulative incidence of NRM at 6 months
  Survival will be tracked during the study, any deaths will be collected. Any death that occurs after hematopoietic stem cell transplantation (HCT) not attributable to relapse of the underlying disease will be considered a non-relapse death.
Cumulative incidence of Non-Relapse Mortality (NRM) at 12 months | 12 months
  Cumulative incidence of NRM at 12 months
  Survival will be tracked during the study, any deaths will be collected. Any death that occurs after HCT not attributable to relapse of the underlying disease will be considered a non-relapse death.
Relapse rate at 6 months | 6 months
  Relapse rate at 6 months
  Relapse, including date of relapse, of the underlying malignancy will be reported.
Relapse rate at 12 months | 12 months
  Relapse rate at 12 months
  Relapse, including date of relapse, of the underlying malignancy will be reported.
Cumulative incidence of chronic GVHD | 12 months
  Cumulative incidence of chronic GVHD requiring systemic steroid treatment by one year from enrollment
Cumulative steroid dose at study day 28 | study day 28
  Cumulative steroid dose at day 28
  Steroid drug and dose is collected weekly for the first 4 weeks of study.
Cumulative steroid dose at study day 90 | study day 90
  Cumulative steroid dose at day 90
  Steroid drug and dose is collected weekly for the first 4 weeks of study, and bi-weekly through study day 90.

CONTACTS AND LOCATIONS:
Overall Officials: John E Levine, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai; Muna Qayed, MD, MS, Principal Investigator — Children's Healthcare of Atlanta, Emory University School of Medicine
Locations (11):
- United States (10):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital Dana Farber Cancer Institute, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin / Children's Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Patient did not consent to this.

DOCUMENTS (1):
  • Informed Consent Form (2023-12-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT05090384/ICF_000.pdf